CLINICAL TRIAL: NCT05913154
Title: A Qualitative Exploration of the Impact of Apathy on the Caregiving Relationship in the Context of Huntington's Disease
Brief Title: Impact of Apathy on Caregiving in HD. Version 1
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of East Anglia (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor
Other Study IDs: 319976
Record Dates: First submitted 2023-05-11; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-03

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cognitive/executive apathy
- Behavioural/inhibition apathy
- Emotional apathy
- Social apathy

SUMMARY:
Huntington's disease (HD) can affect motivation. People with HD may not wash often, keep their house clean and tidy, or eating healthy food. This loss of motivation, or apathy, can also affect the way they talk to people and how willing they are to be in social situations.

There are thought to be four different subtypes of apathy. These include reduced (1) motivation for planning and organising, (2) emotional reactions, (3) thoughts and actions and (4) social interaction.

It is clear from talking to patients and their families in clinic that apathy has a big impact. It is often a source of distress for the people around the patient, who are trying to support and care for them. We know from previous research, that having good social support helps people with Huntington's disease to live independently for longer. This research aims to understand the ways in which apathy can impact the levels of burden felt by caregivers of people with HD.

Caregivers will be asked to take part in a single interview. They will be asked questions about caring for someone with apathy. There will also be the opportunity to share their own first-hand experiences. These interviews will be analysed for common themes using framework analysis. Attention will be given to the relationship between burden and the different types of apathy.

Understanding the factors that lead to increased caregiver burden is the first step towards finding way to support caregivers of people with HD.

ELIGIBILITY:
Inclusion Criteria:

Participants will be included in the study if:

* They hold significant caring responsibilities for someone with clinically manifest HD
* The person they care for scores above the abnormality cut-off determined for HD on one or more subscale of the Dimensional Apathy Scale - Companion version, or the proposed clinical cut-off for the Apathy Motivational Index - Companion.
* They are 18 years or older and able to give valid, informed consent for study participation.

Exclusion Criteria:

Individuals will be excluded from the study is they:

* Have a lack of spoken English, sufficient to affect their understanding of the interview questions or compromise their ability to express their opinions.
* Did not consent to the interview being recorded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Carers of people with Huntington's disease
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Themes | 1 day (Outcomes will be measured once, at the time of the interview)
  Synthesised themes generated from the the qualitative interviews with companions

CONTACTS AND LOCATIONS:
Locations (1):
- University of East Anglia, Norwich, Norfole, United Kingdom